CLINICAL TRIAL: NCT05827289
Title: Pilot Study of the eHealth Application 'Cancer Patients Better Life Experience'
Brief Title: 'Cancer Patients Better Life Experience'
Acronym: CAPABLE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: University of Pavia (Other); University of Haifa (Other); Biomeris s.r.l. (Unknown); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); IBM Research (Unknown); Bitsens JSC (Unknown); Poznań University of Technology (Unknown); Instituti Clinici Scientifici Maugeri (Unknown); Deontics LTD (Unknown); Associazione Italiana Malati di Cancro (Unknown); Universidad Politecnica de Madrid (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P22BLE; NL81970.000.22 (Other: CCMO)
Record Dates: First submitted 2023-01-11; First posted 2023-04-25 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAPABLE cohort (Experimental): Group that receives the CAPABLE application during treatment
  Interventions: Device: Cancer Patients Better Life Experience (CAPABLE)

INTERVENTIONS:
Device: Cancer Patients Better Life Experience (CAPABLE) — The CAPABLE system serves three main goals for the patient: symptom monitoring, information needs fulfilment and interventions to improve mental- and physical wellbeing. These are available to the patient as a smartphone application that is connected to a smartwatch to monitor activity, blood pressure, sleep and heart rate. Patients are able to report symptoms experienced from the treatment and are eligible to do interventions such as mindfulness or yoga. Patients will receive the CAPABLE application and smartwatch for a minimum 3 to a maximum of 6 months after start treatment.

SUMMARY:
The purpose of this study is to compare health-related quality of life, specifically fatigue, in melanoma patients treated with immunotherapy who use or do not use a patient-centered mobile coaching and monitoring system (CAPABLE). It is expected that by using the CAPABLE eHealth tool, patients' fatigue worsens less significantly (10 points) in the first 3 months follow-up than observed in usual care.

DETAILED DESCRIPTION:
This is a prospectively enrolling, explorative cohort study in melanoma patients, eligible for or on treatment with ICI therapy. The explorative cohort receives the CAPABLE smartphone application and a multi-sensorial smartwatch. Patients will be asked to use the system for minimum of three to maximum of six months after enrolment. Questionnaires on health-related quality of life (such as fatigue) and user experience will be administered to the patients on baseline/before start treatment (T0), three months (T1) and six months (T2). Results of this interventional study will be compared with a historical cohort consisting of melanoma patients (P20MEL; NL75996.031.20) with the same inclusion criteria as this study population, but receiving standard care (e.g. without the CAPABLE app).

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Sufficient understanding of the Dutch language
* Participants or their caregiver can use a smartphone (upon patient's consent)
* Histologically confirmed stage III or IV melanoma who receive treatment with immune checkpoint-inhibitors, according to the clinical guidelines.

Exclusion Criteria:

* Included in a clinical trial
* >12 months on active treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue between baseline and 3 and 6 months, as measured by fatigue symptom scale of The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-core 30 (EORTC QLQ-C30) | Baseline, month 3, month 6
  Fatigue is measured on a score from 0-100, the lower the score the less fatigue a patient has

SECONDARY OUTCOMES:
Change in health-related quality of life and QALY's between baseline and 3 and 6 months, as measured by The EuroQoL-5D (EQ-5D-5L). | Baseline, month 3, month 6
  The EQ-5D is a standardised 5-level, 5-dimensional multi-attribute utility questionnaire that measures mobility, self-care, usual activities, pain/discomfort and anxiety/depression. It contains a visual analogue scale, with a score from 0 to 100, the higher the score, the better the outcome. Furthermore, it measures utility scores that can be linked to a country index and be further used in cost-effectiveness analysis.
Change in health-related quality of life and physical symptoms between baseline and 3 and 6 months, as measured by the EORTC QLQ-C30 | Baseline, month 3, month 6
  Funtional domains: scale from 0 to 100, the higher the score, the better the functioning.
  Symptoms: on a scale from 0 to 100, the higher the score, the worse the symptom
Change in melanoma specific quality of life between baseline and 3 and 6 months, as measured by the FACT-M | Baseline, month 3, month 6
  Of the FACT-M, we use the Melanoma Subscale (scale 0 to 64) and the Melanoma Surgery Subscale (scale 0 to 32), items specific to quality of life in melanoma patients. High scores show a high quality of life. The higher the score the better the quality of life is.
Change in patient reported immunotherapy-related toxicity between baseline and 3 and 6 months, as measured by a self-developed questionnaire using EORTC item bank items | Baseline, month 3, month 6
  We identified, based on literature and expert opinion, 19 symptoms and created a symptom list based on items of the EORTC item Library. Scale from 0 to 100, the higher the score, the worse the symptom.
Change in psychological distress between baseline and 6 months, as measured by the Hospital Anxiety and Depression Scale (HADS). | Baseline, month 6
  The HADS is a 14-itemquestionnaire, assesses symptoms of mood disturbance, yielding separate scale scores for anxiety and depression, as well as a total score. The higher the score, the worse the depression and/or anxiety is.
Change in information satisfaction/needs between baseline and 6 months, as measured by the EORTC QLQ-INFO25 | Baseline, month 6
  Measures different domains of satisfaction with delivered information. Scale of 0 to 100, the higher the score the higher the satisfaction/delivered information.
Recruitment rate | Through study completion, an average of 6 months
  The ratio of patients that are included in the study out of the patients eligible for study participation
Patient compliance | Through study completion, an average of 6 months
  The ratio of patients completing the questionnaire and using the CAPABLE app, out of the included patients
Usability/user experience as measured by The System Usability Scale (SUS) | Baseline
  The System Usability Scale (SUS) consists of a 10 item questionnaire with five response options for respondents. The participant's scores are converted to original scores of 0-40 to 0-100. Scores should be considered only in terms of their percentile ranking.
Usability/user experience as measured by PAtient Trust Assessment Tool (PATAT) | Month 3
  Measured on a Likert-scale from 1 to 5. A score higher than 3 is considered trust in telemedicine. Reported as the percentage that has a score higher than 3 and the percentage that scored equal or below 3.
Usability/user experience as measured by the User Version of the Mobile Application Rating Scale (uMARS) | Month 6
  The uMARS is a20-item measure that includes 4 objective quality subscales-engagement, functionality, aesthetics, and information quality-and 1 subjective quality subscale. The higher the score the better the outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Fraterman I, Wollersheim BM, Tibollo V, Glaser SLC, Medlock S, Cornet R, Gabetta M, Gisko V, Barkan E, di Flora N, Glasspool D, Kogan A, Lanzola G, Leizer R, Mallo H, Ottaviano M, Peleg M, van de Poll-Franse LV, Veggiotti N, Sniatala K, Wilk S, Parimbelli E, Quaglini S, Rizzo M, Locati LD, Boekhout A, Sacchi L, Wilgenhof S. An eHealth App (CAPABLE) Providing Symptom Monitoring, Well-Being Interventions, and Educational Material for Patients With Melanoma Treated With Immune Checkpoint Inhibitors: Protocol for an Exploratory Intervention Trial. JMIR Res Protoc. 2023 Oct 11;12:e49252. doi: 10.2196/49252. PMID 37819691